CLINICAL TRIAL: NCT06676189
Title: Comparison of Pivotal Medial Polyethylene Versus Ultra-congruent in Total Knee Arthroplasty
Acronym: MEPCAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2023 DESCAMPS (MEPCAT); 2023-A01565-40 (Other: 2023-A01565-40)
Record Dates: First submitted 2024-10-24; First posted 2024-11-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Replacement; Primary Knee Replacement; Gonarthrosis
Keywords: prospective; randomized study; parallel groups; forgotten joint score
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: Arm 1: Total knee replacement with medial pivot polyethylene
  Arm 2: Total knee replacement with ultra-congruent polyethylene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medial pivot polyethylene (Active Comparator): Total knee replacement with medial pivot polyethylene
  Interventions: Device: total knee arthroplasty with medial pivot polyethylene
- ultra-congruent polyethylene (Active Comparator): Total knee replacement with ultra-congruent polyethylene
  Interventions: Device: total knee arthroplasty with ultra-congruent polyethylene

INTERVENTIONS:
Device: total knee arthroplasty with medial pivot polyethylene — total knee arthroplasty with medial pivot polyethylene
  Arms: medial pivot polyethylene
Device: total knee arthroplasty with ultra-congruent polyethylene — total knee arthroplasty with ultra-congruent polyethylene
  Arms: ultra-congruent polyethylene

SUMMARY:
The aim of this study is to compare the forgotten joint score for the medial pivot polyethylene and ultra-congruent polyethylene which are used in total prosthetic replacement of the knee

DETAILED DESCRIPTION:
Total knee arthroplasty is usually effective at improving the quality of life of patients suffering from arthritis.

Over the years, patient expectations about the quality of life post-implantation continue to rise.

It is therefore essential to improve continuously surgical techniques and implants to fulfill patient expectations in terms of pain and movements.

The prosthetic device is composed of a metallic femoral unit, which imitates the articular surface of the femur, and a metallic tibial baseplate covered with a polyethylene (a highly resistant polymer) insert which articulates between the femur and the tibia. This insert can take several forms such as medial pivot or ultra-congruent.

This polymer provides an interface between the two metallic units forming the prothetic device. It has two roles: it provides a lasting contact surface and it offers stability to the knee in substitution of the ligaments.

In order to achieve this double function, a polyethylene system, called " medial pivot " was conceived.

This system mimics as close as possible the anatomical knee kinematics with a rotational movement that the " ball in socket " tries to reproduce by the mediatisation of the pivot point during knee flexion.

Currently, there are no randomized study which were conducted comparing these two types of polyethylene.

Total knee arthroplasty is usually effective at improving the quality of life of patients suffering from arthritis.

Over the years, patient expectations about the quality of life post-implantation continue to rise.

It is therefore essential to improve continuously surgical techniques and implants to fulfill patient expectations in terms of pain and movements.

The prosthetic device is composed of a metallic femoral unit, which imitates the articular surface of the femur, and a metallic tibial baseplate covered with a polyethylene (a highly resistant polymer) insert which articulates between the femur and the tibia. This insert can take several forms such as medial pivot or ultra-congruent.

This polymer provides an interface between the two metallic units forming the prothetic device. It has two roles: it provides a lasting contact surface and it offers stability to the knee in substitution of the ligaments.

In order to achieve this double function, a polyethylene system, called " medial pivot " was conceived.

This system mimics as close as possible the anatomical knee kinematics with a rotational movement that the " ball in socket " tries to reproduce by the mediatisation of the pivot point during knee flexion.

Currently, there are no randomized study which were conducted comparing these two types of polyethylene.

ELIGIBILITY:
Inclusion criteria :

* Subjects 18 to 90 years of age, eligible for a primary total knee replacement for gonarthrosis
* Competent subjects able to give informed consent to participate in the research
* Affiliation to the social security system

Exclusion criteria :

* Infection history of the knee to be replaced
* Deformity greater than 15 degrees
* Any surgical and/or anesthetic contraindication, or any condition deemed by the investigator to be incompatible with the research.
* Any contraindication mentioned in the instructions for use of the medical device
* Pregnant or breastfeeding women
* Recent infection history of the surgical site
* Adults who are subject to a legal protection measure or who are unable to express their constent (Article L1121-8 of the French Public Health Code) and subjects under judicial protection (article L. 1122-2 FPHC)
* Subjects who refuse to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
evaluation of the forgotten joint score (FJS12) | Day 45
  Forgotten knee score at 6 weeks (FJS-12, evaluated out of 100), which allows the analysis of quality of life specifically in relation to knee pathologies
evaluation of the forgotten joint score (FJS12) | Month 12
  Forgotten knee score at 6 weeks (FJS-12, evaluated out of 100), which allows the analysis of quality of life specifically in relation to knee pathologies

SECONDARY OUTCOMES:
knee joint mobility | Day -1
  Measurement of mobility in degrees (scale from 0 to 10)
knee joint mobility | Day 45
  Measurement of mobility in degrees (scale from 0 to 10)
knee joint mobility | month 12
  Measurement of mobility in degrees (scale from 0 to 10)
pain assessment | Day -1
  assessment with a numeric pain rating scale ranging from 0 (none) to 10 (severe pain)
pain assessment | day 45
  assessment with a numeric pain rating scale ranging from 0 (none) to 10 (severe pain)
pain assessment | month 12
  assessment with a numeric pain rating scale ranging from 0 (none) to 10 (severe pain)
the Knee Society Score (KSS) | Day -1
  the KSS (free of charge) scoring system is divided into 2 subcategories: a clinical score (maximum of 100 points) and a functional score (maximum of 100 points)
the Knee Society Score (KSS) | Day 45
  the KSS (free of charge) scoring system is divided into 2 subcategories: a clinical score (maximum of 100 points) and a functional score (maximum of 100 points)
the Knee Society Score (KSS) | month 12
  the KSS (free of charge) scoring system is divided into 2 subcategories: a clinical score (maximum of 100 points) and a functional score (maximum of 100 points)
Knee injury and Osteoarthritis Outcome Score Physical Function Short form (KOOS-PS). | day -1
  the KOOS-PS (free of charge) is used to assess the postoperative quality of life related to knee joint pathologies.
Knee injury and Osteoarthritis Outcome Score Physical Function Short form (KOOS-PS). | Day 45
  the KOOS-PS (free of charge) is used to assess the postoperative quality of life related to knee joint pathologies.
Knee injury and Osteoarthritis Outcome Score Physical Function Short form (KOOS-PS). | Month 12
  the KOOS-PS (free of charge) is used to assess the postoperative quality of life related to knee joint pathologies.
radiographic alignment | month 12
  measurement of the anteroposterior radiographic alignment at 1 year post-operative using the Hip-knee-ankle (HKA) angle
radiological complications | Day -1
  Peri- and post-operative complications using standard radiographic analysis (static radiographs of the lower limbs, anteroposterior and lateral knee radiographs, patellofemoral view at 45°)
radiological complications | Day 45
  Peri- and post-operative complications using standard radiographic analysis (static radiographs of the lower limbs, anteroposterior and lateral knee radiographs, patellofemoral view at 45°)
radiological complications | Month 12
  Peri- and post-operative complications using standard radiographic analysis (static radiographs of the lower limbs, anteroposterior and lateral knee radiographs, patellofemoral view at 45°)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DESCAMPS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No